CLINICAL TRIAL: NCT06713213
Title: Clinical Comparison of FRNDS Cannula and Plethysmography Belts
Brief Title: Clinical Comparison of Flow Regulated Nasal Oxygen Delivery System (FRNDS) Cannula and Plethysmography Belts
Acronym: FRNDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB # 24-813; HRPP Protocol 24-813 (Other: Carilion Innovations, Virginia Tech University)
Record Dates: First submitted 2024-09-20; First posted 2024-12-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Failure With Hypoxia

STUDY DESIGN:
Intervention Model Description: INTERVENTIONS:
  * RIP belts will be calibrated and outfitted on participants chests during each visit. RIP belts will be stored on-site and will be calibrated and outfitted by a designated member of the study
  * FRNDS cannulas will be placed inside nasal cavity, identical to clinical practices. FRNDS cannulas will be transported between the two sites according to participant enrollment
  * Digital calipers to measure both vertical and horizontal dimensions of the nasal cavity 1cm from the opening. Calipers will be appropriately cleaned before and after each use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concomitant comparison of respiratory volumes using FRNDS device with Plethysmography belts (Experimental): FRNDS is a novel cannula device that can both measure tidal volume (VT) in real time while simultaneously delivering air to the patient.
  Study subjects with undergo continuous measurement of a patient's VT while simultaneously delivering variable volumes of air to the patient and comparing these results with VTs captured with conventional technology (RIP belts)
  Interventions: Other: Flow-regulated nasal oxygen delivery system (FRNDS)

INTERVENTIONS:
Other: Flow-regulated nasal oxygen delivery system (FRNDS) — FRNDS is a novel cannula device that can both measure tidal volume (VT) in real time while simultaneously delivering air to the test subject.
  After collecting data without any flow through the FRNDS cannula for 2 minutes, varying amounts of medical air ( 21% Fio2) starting with 2 Liters for two minutes , 4 liters for 2 minutes, 6 liters for two minutes and 8 liters for two minutes would be delivered while monitoring and recording data previously described with the FRNDS device.

SUMMARY:
SUMMARY:

This is a quantitative, non-inferiority study using healthy participants to compare tidal volumes at rest measured by both a standard RIP belt and a flow-regulated nasal oxygen delivery system FRNDS cannula.

Recording of tidal breathing is essential for patients undergoing evaluation for respiratory disease and reduced exercise capacity. Conventional spirometry techniques involving pneumotachometers are currently employed worldwide in pulmonary testing laboratories to record pulmonary flow and calculate tidal volumes by allowing subjects to breath out of mouth into these devices. However, concurrent use of pneumotachometers while testing a novel nasal device is not feasible. Respiratory inductive plethysmography (RIP) has been developed and validated to evaluate tidal ventilation during quiet breathing using a band around the chest. RIP signals may be contaminated by body movements resulting in artifacts which may be a limitation. However, although a crude method when compared to spirometry, RIP remains a viable method for comparison.

FRNDS is a novel cannula device that can both measure tidal volume (VT) in real time while simultaneously delivering air to the patient. The gold-standard of measuring VT clinically is spirometry; however, this test cannot be completed when patients are receiving supplemental oxygen or air.

Thus far, the FRNDS cannula has been tested in vitro with a cylindrical flow model and has accurately measured simulated VTs with 80% accuracy, but has not yet been validated in Human subjects. To assess the devices robustness in a clinical scenario is essential to the development and eventually adaptation of FRNDS in clinical care.

OBJECTIVES:-

In this study the investigators aim to describe and validate flow-regulated nasal oxygen delivery system (FRNDS) instrumented nasal cannula as a non-inferior methodology of measuring flows at the nasal interface compared to conventional methods (e.g., RIP belts) with the added benefit of administering a dose of air to the subjects.

While the FRNDS device was validated in vitro in a cylindrical model, the investigators aim to show equivalence to standard respiratory measurement methods in healthy subjects. This milestone will be essential towards the eventual translation of an adaptive cannula system that measures and adjusts air flow according to patient needs in real time.

ENDPOINTS:

The primary endpoint of this study is the continuous measurement of a test subjects Vt and Minute ventilation ( VE) while simultaneously delivering variable volumes of air to the patient and comparing these results with Vts and VE captured with conventional technology (RIP belts). The investigators will also be collecting inspiratory time (Ti) expiratory time (Te) continuously and a single measurement of nasal cavity openings (e.g., internal vertical and horizontal dimensions 1 cm inside the nares using calipers)

DETAILED DESCRIPTION:
STUDY DESIGN:

For each subject, over the 10-minute period the investigators will be collecting time-series data consisting of tidal volume (VT, VE derived from a fluid dynamics modeling equation based on pressure sensors and the measured diameter of the patient & nasal cavity), inspiratory time (Ti), and expiratory time (Te). Accordingly, minute ventilation will be calculated throughout the trial. Mean, standard deviation, and quartile (e.g., 25th, 50th, and 75th) measurements will be calculated after the trial is complete.

In addition, using the aforementioned measurements and the nasal cavity diameter measurements taken at the beginning of the trial, the investigators will be comparing the accuracy of the VT derived from our measure nasal cavity diameters and compare them to statistical nasal cavity sizes based on participant demographics (Corey et al. Otolayngol Head Neck Surg 1998; 119:389-93). Means, standard deviations, and quartile measurements will be compared between the measured and statistical nasal cavity diameter groups.

The data collected from RIP belts and the FRNDS cannula will be measured via descriptive statistics (e.g., mean, variance, standard deviation), a paired t-Test, Cross-Correlation Function, mean squared error (to determine absolute differences between measurements), and potentially dynamic time warping (DTW) to account for shifts and distortions in time.

METHODOLOGY:

All data collected during each trial is considered minimally invasive and poses a non-significant risk to subjects.

1. Participant Outreach and Screening 1.1 Via email or the QR code provided on the flyer, potential subjects will receive a quick screening tool as outlined in FRNDS_study_screening questionnaire. If no contraindications are found, participants will be forwarded to a calendar with potential study times. These forms will be filled out without the collection of names.

   1.2 Subjects will receive a downloadable calendar invite for their designated time and a copy of the consent form for review prior to their appointment. If cancelation or rescheduling is required, subjects are encouraged to email adogan@vt.edu stating their original timeslot.

   1.3 Subjects who walk in; for a study time will be verbally asked the questions outlined in the FRNDS_study_screening questionnaire, and if no contraindications are found, will be consented and trialed without an appointment.
2. Subjects Consenting and Questionnaire 2.1 At the time of study participation, study investigators for that time will go over the information outlined in the consent form.

   2.2 Consented subjects will fill out the questionnaire outlined in the FRNDS_study_questionnaire. If for some reason any exclusion criteria are met, participants will be informed they are unable to participate and will not be eligible for the gift card. At this time, participants will be assigned a number in the format of (Location-Date-Time-Participant Number) (for example: SIM-09082024-1445-2)
3. Nasal Cavity Measurements 3.1 Digital calipers will be used to measure vertical and horizontal diameters of the nasal cavity. Digital calipers will be cleaned and disinfected using alcohol wipes between each use.
4. FRNDS cannula and RIP belt measurements 4.1 Subjects will be seated comfortably on a chair and be outfitted by investigators with the RIP belt along their chest and the cannula under their nose. RIP belts will be briefly calibrated based on participant body habitus by monitoring passive breathing and 1-2 full, deep breaths. Each subject will receive a new cannula, which is tested prior to each trial for leakage.

4.2 Participants will then be measured according to the previously described protocol. A video recorded will be started pointing at the RIP belt analog output for timestamping.

4.2.1 2 minutes of data collection on room air at atmospheric pressure 4.2.2 2 minutes of data collection on 2L room air 4.2.3 2 minutes of data collection on 4L room air 4.2.4 2 minutes of data collection on 6L room air 4.2.5 2 minutes of data collection on 8L room air

5. Study conclusion 5.1 RIP belts and cannula will be removed from participants 5.2 If requested, participants can see and record their cannula results on-site

DATA COLLECTION

Subjects with histories of chronic lung disease, chronic heart disease, neuromuscular disease, nasal surgery, deviated nasal septum, or exclusive mouth breathers will be excluded from this study. Subjects that meet exclusion criteria during the questionnaire will be excluded from the study and will not be eligible for gift card compensation.

Subjects will be seated comfortably and will be at-rest for the duration of the study.

Subjects will have full ability to withdraw from the study at any time. Any equipment including calipers used for multiple participants will be disinfected with alcohol wipes to avoid contamination between subjects. Each subject will receive a new cannula, which is checked before each trial.

Data will be collected using the following methods:

1. FRDNS_study_screening, which is given prior to consent and does not include identifiable information. This information will not be stored and only acts as a filter before subjects can book time slots (e.g., only participants who do not meet exclusion criteria will be directed to time slot booking page)
2. FRNDS_study_questionnaire which is given after subject consent. This information will only be organized based on site location, date and time and this information will be used in analysis.
3. RIP belt monitoring. Analog output from the RIP belt during the study will be recorded via video for timestamping. The video will not have audio and will only show analog output from the belt.
4. FRNDS cannula output. Digital output from the cannula will be sent to a local onsite computer and will be identified with the same Participant ID as outlined in the FRNDS_study_questionnaire, which will be manually inputted by study investigator

   Emails will only be obtained by subjects who cancel or reschedule their study time slots, but this information will not be included in the final study.

   Names and signatures will be collected on the consent form prior to any analyzable data collection.

   Ti, Te and VT/VE will be collected by RIP belts and FRNDS cannulas simultaneously, non-invasively. Briefly, RIP belts measure the physical displacement and pressure generated by the participants chest during inhalation and exhalation. The FRNDS utilizes pressure sensors embedded within the device to derive air flows and inhale/exhale times. These will be identified via Subject ID, as previously described.

   Basic demographic information (e.g., age, gender, height, weight, and race) will be collected along with basic health information according to inclusion/exclusion criteria (see the FRNDS_study_questionnaire document for exhaustive list of questions) No identifiable personal health information will be gathered, participants will be identified with a unique Participant ID as previously described.

   Nose cavity diameters will be collected on-site before beginning each trial. This will also be matched according to Subject ID.

   SAFETY AND OVERSIGHT:

   RIP belts (Brand: Respirate) will be used to measure VT of participants at rest. Use will not deviate from FDA-approved usage.

   FRNDS cannula will also be used to measure VT of participants at rest. Use will not deviate from the clinical administration of a standard nasal cannula. FRNDS cannula will be connected to a standard air delivery system including an air-oxygen mixer, flow meter, and an active humidifier/heater to create a complete breathing circuit.

   The FRNDS cannula is not currently FDA-approved; however, based on our assessment, the investigators have determined that the device qualifies as a non-significant risk (NSR) device, and therefore, it is exempt from the requirement for an Investigational Device Exemption (IDE). This determination is based on the following specific considerations:
   * Non-invasive Nature:

   The FRNDS cannula is a non-invasive device, identical in form and function to standard FDA-approved nasal cannulas that are widely used for delivering air or supplemental oxygen. It does not penetrate the body or pose any risk to tissue, organ systems, or other bodily functions.

   -- Interaction with the Subject: The novel components of the FRNDS system, such as the pressure sensors, do not directly interact with the participant. These sensors are solely connected to the air-delivery cannula and are used only to monitor airflow and pressure changes within the tube itself. No electrical components or novel circuits have any direct contact with the participant, ensuring there is no additional risk beyond what is posed by a standard cannula.

   -- Use of Room Air: The FRNDS device delivers room air, not supplemental oxygen, further reducing any respiratory or fire-related risks that may be associated with devices delivering oxygen-enriched air.
   * Established Device Foundation:

   The cannula itself is based on FDA-approved, off-the-shelf components (e.g., Fisher & Paykel high-flow cannulas), and minimal modifications have been made to the cannula that would not alter its interaction or delivery of air to the subject.

   -- Comparable Risks to Standard Care: The risks associated with the FRNDS cannula are no greater than those encountered with standard nasal cannulas that are routinely used in clinical settings for the delivery of room air or supplemental oxygen. As such, the risks posed are minimal and consistent with everyday clinical practice.

   -- Minimal Risk to Participants: Given the non-invasive nature of the device and the absence of direct interaction between the patient and the novel components, the FRNDS device is classified as posing no significant risk (NSR) to subjects. This aligns with the FDAs definition of an NSR device, which includes devices that present minimal risk comparable to those encountered in daily life or during routine clinical evaluations.

   In conclusion, the investigators affirm that the FRNDS device qualifies for a non-significant risk determination, exempting it from the IDE requirement.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy adults over the age of 18.

Exclusion Criteria:

* Adults with preexisting comorbidities including:
* Chronic lung disease
* Chronic heart disease
* Neuromuscular disease
* History of nasal surgery
* History of upper airway reconstructive surgery
* History of deviated nasal septum
* Preferential mouth breathers
* Minors, as defined by state law where the study is performed (infants, children, teenagers)
* Pregnant women will be excluded, as they have physiologically altered respiratory parameters and to minimize potential mechanical discomfort due to the RIP belts.
* Prisoners (including all incarcerated individuals)
* Adults not capable to consent on their own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Tidal volumes ( Minute Ventilation) and comparison of novel device with standard technology | Through study completion, an average of 1 year.
  Continuous measurement of a patients VT and Minute Ventilation while simultaneously delivering variable volumes of air to the subjects and comparing these results with VTs and Minute ventilation captured with conventional technology (RIP belts)

SECONDARY OUTCOMES:
Continuous measurement of Inspiratory time (Ti), and expiratory time (Te) and minute ventilation and comparison with standard technology | Through study completion, an average of 1 year.

OTHER OUTCOMES:
Comparison of tidal volume from nasal cavity diameter with statistical nasal cavity sizes | Through study completion, an average of 1 year.
  Comparing the accuracy of the VT derived from our measure nasal cavity diameters and compare them to statistical nasal cavity sizes based on participant demographics

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Carilion Clinic Center for Simulation, Research and Patient Safety, Roanoke, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No
Since this clinical trial is designed to test and validate the prototype in healthy human subjects, the investigators would like to exercise discretion and prevent disseminating information that my compromise the intellectual property.

REFERENCES:
- [Background] Girardis M, Busani S, Damiani E, Donati A, Rinaldi L, Marudi A, Morelli A, Antonelli M, Singer M. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1583-1589. doi: 10.1001/jama.2016.11993. PMID 27706466
- [Background] Agusti A, Vogelmeier CF. GOLD 2024: a brief overview of key changes. J Bras Pneumol. 2023 Dec 22;49(6):e20230369. doi: 10.36416/1806-3756/e20230369. No abstract available. PMID 38126685
- [Background] Stevenson NJ, Walker PP, Costello RW, Calverley PM. Lung mechanics and dyspnea during exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1510-6. doi: 10.1164/rccm.200504-595OC. Epub 2005 Sep 15. PMID 16166620
- [Background] Alobaidi NY, Stockley JA, Stockley RA, Sapey E. An overview of exacerbations of chronic obstructive pulmonary disease: Can tests of small airways' function guide diagnosis and management? Ann Thorac Med. 2020 Apr-Jun;15(2):54-63. doi: 10.4103/atm.ATM_323_19. Epub 2020 Apr 3. PMID 32489439
- See also: Lamb K, Theodore D, Bhutta BS. Spirometry. [Updated 2023 Aug 17]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2024 Jan-. — https://www.ncbi.nlm.nih.gov/books/NBK560526/
- See also: Torp KD, Modi P, Pollard EJ, Simon LV. Pulse Oximetry. 2023 Jul 30. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2024 Jan-. PMID: 29262014. — https://www.ncbi.nlm.nih.gov/books/NBK470348/
- See also: Pulse Oximetry Klaus D. Torp; Pranav Modi; Elizabeth J. Pollard; Leslie V. Simon. — https://www.ncbi.nlm.nih.gov/books/NBK470348/